CLINICAL TRIAL: NCT05691166
Title: Reducing Falls With Progressive Resistance Training (ReFit) for the Oldest Old Adults With Sarcopenia. A 12-month Randomised Controlled Trial (RCT).
Brief Title: Reducing Falls With Progressive Resistance Training for the Oldest Old Adults With Sarcopenia
Acronym: ReFit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022/462261
Record Dates: First submitted 2022-12-16; First posted 2023-01-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Aging
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive resistance training (Experimental): Twice weekly high-intensity progressive resistance training for 12 months
  Interventions: Behavioral: High-intensity progressive resistance training
- Control (Active Comparator): Participants randomised to the control group receive a booklet containing Norway's current recommendations for physical activity for older adults. These recommendations mean ≥150 minutes of moderate-intensity or ≥75 minutes of vigorous-intensity physical activity per week and two to three weekly balance and resistance training sessions. The booklet also includes pictures and instructions for seven exercises to help prevent falls.
  Interventions: Other: General practitioner care

INTERVENTIONS:
Behavioral: High-intensity progressive resistance training — Supervised high-intensity progressive resistance training twice per week for 12 months
  Arms: Progressive resistance training
Other: General practitioner care — Referred to general practitioner (GP) for further follow-up. The GPs will be informed about participants sarcopenia status with results from assessments of muscle strength, muscle mass, and physical performance. The management of the sarcopenia is at the GPs own discretion.
  Arms: Control

SUMMARY:
This study will investigate the effects of 12 months of high-intensity progressive resistance training compared with a control group on fall-rate in older adults with sarcopenia.

DETAILED DESCRIPTION:
Despite the wealth of theoretical benefits, existing literature on resistance training for falls prevention is not conclusive, given the sub-optimal resistance training paradigms, poor study quality, and use of multimodal training interventions, precluding isolation of the resistance training benefits. It is also possible that resistance training benefits for falls reduction will be most evident in those with sarcopenia to begin with as a risk factor for their falls. We will therefore conduct a randomised, controlled trial assessing the effects of resistance training reduce falls in the oldest old adults with sarcopenia, as well as to increase strength and muscle mass.

Amendment 2023-12-15: The description of the control condition was updated following ethics committee approval. Referral to the general practitioner for follow-up was replaced with provision of written information on current physical activity recommendations for older adults. This change was made to improve acceptability and feasibility of the control condition; the study outcomes and intervention were unchanged.

Amendments: 2024-09-18. We updated the low grip-strength inclusion criterion from [Men:<39.6kg, Women:<21.4kg] to [Men:<41.6kg, Women:23.4kg] based on normative values (Ref: Svinøy, O. E., Hilde, G., Bergland, A., & Strand, B. H. [2023]).

Extension amendment (2025-09-02): With new funding and ethics approval (REK 2022/462261), we added post-trial follow-up at 24 and 36 months to evaluate disability-free survival and the durability of effects on falls and several secondary outcomes. Falls during follow-up are collected via 12-month recall. No changes to interventions or the prespecified 0-12-month primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Aged 80 years or older
* Low muscular strength (grip strength: <41.3 kg for males and <23.4 kg for females [from 18.09.2024] or chair stand >15 seconds)
* Community-dwelling incl. independent senior housing
* Ambulatory without supervision or physical assistance from another person. Assistive devices such as canes/crutches/walkers allowed.
* Able to see and hear sufficiently to undertake assessments and partake in the planned exercise training.

Exclusion Criteria:

* Pre-existing diagnosis of dementia
* Moderate or severe cognitive impairment (score <18 on the Mini-Mental State Examination)
* Living in institutional care
* Non-ambulatory or requiring person or wheelchair to assist when walking
* Degenerative neurological and neuromuscular disease/disorder significantly influencing gait and mobility (e.g. amyotrophic lateral sclerosis [ALS] and Parkinson's disease).
* Amputation (other than toes)
* Contraindications to resistance training
* Unstable fracture
* Inability to comply with study requirements
* Currently undertaking progressive resistance training

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Falls | 12 months
  Relative risk for falls, fall rate per person years. Self-report.

SECONDARY OUTCOMES:
Falls | 6 months
  Relative risk for falls, fall rate per person years. Self-report.
Falls | 6, 12, 24, and 36 months.
  Number of falls, number of fallers/nonfallers/frequent fallers, and time to first fall. Self-report.
Falls requiring medical attention | 6, 12, 24, 36 months
  Number of falls requiring medical attention. Collected via self-report and ascertained by linkage to the Norwegian Patient Registry and medical journals with the use of unique 11-digit Norwegian national identification number for each participant.
Fall-related injuries | 6, 12, 24, 36 months
  Classified according to the International Classification of Diseases, 11th revision, classification system. Peripheral fracture rate per person-years, number of peripheral fractures, number of people sustaining peripheral fractures, and number of people sustaining multiple events. Collected via self-report and ascertained by linkage to the Norwegian Patient Registry and medical journals with the use of unique 11-digit Norwegian national identification number for each participant.
Dynamic muscular strength | 6 and 12 months
  1-repetition maximum leg press and leg extension
Grip strength | 6, 12, 24, 36 months
  Maximal isometric handgrip strength
Muscular power | 6 and 12 months
  Muscular power assessed using a force platform installed on a leg press machine
Physical performance | 6, 12, 24, 36 months
  Physical performance using the Short Physical Performance Battery
Balance | 6, 12, 24, 36 months
  Static and dynamic balance using the Mini-Balance Evaluation Systems Test (BESTest)
Stature | 6, 12, 24, 36 months
  Stretch stature using a wall-mounted stadiometer
Body mass | 6, 12, 24, 36 months
  Body mass estimated using multi-frequency bioelectrical impedance analysis
Body composition | 6, 12, 24, 36 months
  Estimated using multi-frequency bioelectrical impedance analysis. Fat mass, skeletal muscle mss, appendicular skeletal muscle mass.
Circumferences | 6 and 12 months
  Waist, arm, and calf circumference
Resting blood pressure and resting heart rate | 6, 12, 24, 36 months
  Systolic and diastolic blood pressure, and resting heart rate measured after 5 minutes of seated resting using an automated blood pressure device
Orthostatic blood pressure | 6, 12, 24, 36 months
  Systolic and diastolic blood pressure response 1, and 3-min after standing up
Physical activity | 6, 12, 24, 36 months
  Self-reported physical activity levels
Health-related quality of life | 6, 12, 24, 36 months
  Health-related quality of life assessed using the 12-item Short-form health survey
Fear of falling | 6, 12, 24, 36 months
  Fear of falling assessed using the Falls Efficacy Scale-International
Cognitive function | 6 and 12 months
  Cognitive function evaluated using The Mini Mental State Examination
Depression | 6, 12, 24, 36 months
  Levels of depression measured via the Geriatric Depression Scale.
Frailty | 6, 12, 24, 36 months
  Physical frailty assessed according to Fried's frailty phenotype
Nutritional status | 6, 12, 24, 36 months
  Nutritional status assessed using the Mini-nutritional Assessment Short form.
Sleep quality | 6, 12, 24, 36 months
  Sleep quality assessed using the Pittsburgh Sleep Quality Index
Hospital admissions | 0-12 months and 0-36 months
  Information about hospitalisations due to falls and fall-related injuries will be collected by means of electronic linkage to the Norwegian Patient Registry and medical journals with the use of a unique 11-digit Norwegian national identification number for each participant.
Use of primary health care, community care, and assistive technology | 0-12 months and 0-36 months
  Use of primary health care (general practitioner, emergency room, physiotherapist, and chiropractor), community care, and assistive technology during the study will be collected by linkage to the Norwegian Municipal Patient and User Register (KPR) database with the use of a unique 11-digit Norwegian national identification number for each participant.
Use of prescription drugs | 12 months
  Use of prescription drugs during the study will be collected by linkage to the Norwegian Prescribed Drug Registry with the use of a unique 11-digit Norwegian national identification number for each participant.
Disability-free survival (DFS) | Baseline to 36 months post-randomisation
  DFS is defined as time from randomization to the first occurrence of: (i) death from any cause; (ii) incident dementia; or (iii) incident ADL disability. Participants with dementia or ADL disability at baseline are excluded from the DFS analysis.
  Death: ascertained by linkage to the Norwegian Cause of Death Registry.
  Incident ADL disability: score of 3-5 any of the six primary ADLs (Physical Self-Maintenance Scale) or a score of 0 for any of the five instrumental ADLs (Lawton IADL Scale). If ADL status cannot be obtained, admission to long-term nursing care (national registries) will be used as a proxy for disability.
  Incident dementia: registry/clinical diagnosis (ICD-10 F00-F03, G30, or equivalent codes in national registries). Exploratory supplement: MoCA assessed at 24/36 months; dementia defined as MoCA z-score ≤ -2.0 (age/education-adjusted).
Healthcare and implementation costs | 0-12 months
  Intervention costs (resistance training and control), prescription medication, and health and care service utilisation during the 12-month intervention period. Costs for the training intervention include fitness centre membership fees and instructor labour costs (time worked + overheads). We will not consider potential travel costs for participants. We will obtain expenses related to prescription medication and health care service utilisation by linking participant data with data from the Norwegian Prescribed Drug Registry, the Norwegian Patient Registry (specialist health services), and the Municipal Patient and User Register (primary care, care services, physiotherapist, and chiropractor). We focus only on implementation costs, thus disregarding research protocol costs (e.g. recruitment).
Quality-Adjusted Life-Years (QALY's) | 0-12 months
  We use the 12-item short-form health survey (SF-12) to assess health-related quality of life across eight areas, with scores summed into a physical component summary score and a mental component summary score, ranging from 0 to 100, with higher scores indicating a better quality of life.32 Next, we'll convert the SF-12 scores into SF-6D utility scores using the equation by Brazier and Roberts (2004).33 The utility scores range from 0 (equivalent to death) to 1 (equivalent to perfect health). Finally, we'll calculate QALYs for the 12-month intervention period by linearly interpolating SF-6D utility scores for baseline, six, and 12 months

OTHER OUTCOMES:
Musculoskeletal pain | 6 and 12 months
  Musculoskeletal pain assessed using the "yes" or "no" question, "during the last year have you had pain in your muscles and/or joints that lasted for at least 3 consecutive months?". When answering "yes", participants will be asked to indicate the affected body areas. In addition, we will assess pain intensity for lower back and neck, specifically, using a 10-cm visual analogue scale (VAS).
Changes in cardiac structure and function | 12 months
  Echocardiographic indices of atrial and ventricular structure and function
Mortality | 0-12 and 0-36 months
  During the study unreported mortality will be assessed twice per year by linkage to the Norwegian population registry with the use of a unique 11-digit Norwegian national identification number for each participant.
Cognitive function | 24 and 36 months
  Montreal Cognitive Assessment Tool
Protein intake | 12, 24, 36 months
  Using the Protein Screener 55+
Incremental cost-effectiveness ratio (ICER) | 0-12 months
  We will analyse the cost-effectiveness by estimating the Incremental Cost-Effectiveness Ratio (ICER) between the resistance training and control groups. We consider resistance training cost-effective if the ICER falls below the willingness-to-pay threshold (WTP).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berg, PhD, Principal Investigator — Norwegian University of Science and Technology; Øivind Rognmo, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway